CLINICAL TRIAL: NCT02042781
Title: An Open-label, Multi-centre Phase I Study of the Safety and Tolerability of IV Infused PG545 in Patients With Advanced Solid Tumours
Brief Title: Study of the Safety and Tolerability of IV Infused PG545 in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zucero Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG545102
Record Dates: First submitted 2014-01-14; First posted 2014-01-23 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Advanced Solid Tumours
Keywords: PG545; Phase I; Progen; antimetastatic; antiangiogenic; advanced cancer patients; solid tumors; solid tumours; tumor microenvironment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PG545 (Experimental): Once weekly, one hour IV infusion of PG545.
  Interventions: Drug: PG545

INTERVENTIONS:
Drug: PG545 — PG545 will be administered once weekly, as a one hour IV infusion. Patients will be treated until they exhibit disease progression, withdraw due to poor tolerability, or the study reaches its defined end-point. This study is a dose escalation study with doses of 25 mg to 250 mg anticipated.

SUMMARY:
This Phase Ia study aims to establish the maximum tolerated dose of once-weekly IV infused PG545 and to evaluate its safety in subjects with advanced solid tumours. In addition, the study will explore whether PG545 exposure results in changes to chemicals produced by the body that are associated with cancer growth and spread.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years.
* Histological or cytological documentation of non hematologic, malignant solid tumour.
* Have failed at least one previous therapeutic regimen.
* LIfe expectancy >= 12 weeks.
* ECOG performance status 0 or 1.
* Written, signed and dated informed consent.
* Able and willing to meet all protocol-required treatments, investigations and visits.
* Have adequate organ function.

Exclusion Criteria:

* Clinically significant non-malignant disease.
* Active CNS metastases.
* Subjects with uncontrolled diabetes.
* History of clinically significant adverse drug reaction to heparin or other anti-coagulant agents
* Concomitant use of aspirin (> 150 mg/day), NSAIDs (except COX-2 selective inhibitors), vitamin K antagonists (other than low-dose), heparin within two weeks prior to randomisation, or other anti-platelet drugs.
* History of severe allergic, anaphylactic or other significant adverse reaction to radiographic contrast media.
* Known seropositivity to the human immunodeficiency vies (HIV)
* Women who are pregnant or breast feeding
* Women of child-bearing potential and male subjects who are partners of women of child bearing potential who are unable or unwilling to use effective means of contraception.
* Subjects who have received an investigational agent within 28 days prior to Cycle 1 Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-01; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Determination of maximum tolerated dose (MTD) of PG545 | Evaluated at the end of initial 28-day cycle
  The MTD will be determined by assessing dose limiting toxicities at the end of the first month's treatment. Dose escalation and de-escalation will continue until an MTD is identified. Each cohort of patients will receive weekly doses at a single dose level for the duration of the study.

SECONDARY OUTCOMES:
Number of adverse events by cohort | Subjects will be followed for the duration of their treatment (an expected average of 12 weeks), and for four weeks post-treatment
Severity of adverse events by cohort | Subjects will be followed for the duration of their treatment (an expected average of 12 weeks), and for four weeks post-treatment
Assessment of the anti-tumour activity of PG545 using RECIST criteria | Subjects will be followed for the duration of their treatment (an expected average of 12 weeks), and then up to four weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Millward, MBBS, Principal Investigator — Sir Charles Gairdner Hospital
Locations (2):
- Australia (2):
  - Nucleus Network Ltd, Melbourne, Victoria
  - Linear Clinical Research Ltd, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hammond E, Haynes NM, Cullinane C, Brennan TV, Bampton D, Handley P, Karoli T, Lanksheer F, Lin L, Yang Y, Dredge K. Immunomodulatory activities of pixatimod: emerging nonclinical and clinical data, and its potential utility in combination with PD-1 inhibitors. J Immunother Cancer. 2018 Jun 14;6(1):54. doi: 10.1186/s40425-018-0363-5. PMID 29898788